CLINICAL TRIAL: NCT01872676
Title: Immediate Effects of Upper Thoracic Manipulation on Skin Surface Temperature of T3 Vertebral Region and Biceps Brachii Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Amanda Carine Packer, Amanda Carine Packer, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1144-0316
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Myofascial Dysfunction
Keywords: Thermography; Skin Temperature; Manipulation, Spinal; Physical Therapy Modalities
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulation (Experimental): The experimental group received upper thoracic manipulation of the T3 vertebra. The volunteer was instructed to lie in the supine position, interlace her fingers and position her hands in the posterior region of the base of the neck. The therapist than positioned a stabilizing hand in a pistol grip immediately caudal to the T3 vertebra, pushing the volunteer's arms downward to generate flexion of the upper thoracic spine.
  Interventions: Other: Spine manipulation
- Sham (Sham Comparator): The placebo group was placed precisely as the experimental group, with the exception of the positioning of the therapist's hand, which remained with the palm open and not in a pistol grip. Once positioned, the volunteers were instructed to breathe deeply. The maneuver was terminated after one cycle of deep breathing.
  Interventions: Other: Manipulation sham

INTERVENTIONS:
Other: Spine manipulation
  Arms: Manipulation
Other: Manipulation sham
  Arms: Sham

SUMMARY:
The aim of the present study was to assess the immediate effects of upper thoracic manipulation on skin surface temperature in the region of the T3 vertebra and biceps brachii muscle in healthy women. It is a randomized controlled blind study. Twenty-six healthy women of the university community were randomly allocated to an experimental group (n = 13) and a placebo group (n = 13). A single session of the upper thoracic spine manipulation (segment T3)was performed. Infrared thermography was used to determine changes in skin surface temperature in the region of T3 and the biceps brachii muscle, which would indirectly reflect sympathetic activity. Images were taken prior to manipulation, immediately after and both five and 10 minutes after manipulation. Repeated measures ANOVA with the post hoc Bonferroni test and the independent samples t-test were used for the intragroup and intergroup comparisons, respectively, with the level of significance set to 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* 18 and 30 years of age

Exclusion Criteria:

* use of vasoactive medication
* body mass index greater than 25 kg/m2
* having undergone spinal manipulation in previous month
* and any red flag sign, such as malignant tumor, inflammatory or infectious disease that contraindicated manual therapy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Skin temperature | 1 years
  Infrared thermography was used to determine changes in skin surface temperature in the region of T3 and the biceps brachii muscle, which would indirectly reflect sympathetic activity. Images were taken prior to manipulation, immediately after and both five and 10 minutes after manipulation.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Packer, MSc, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Methodist University of Piracicaba, Piracicaba, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.unimep.br/